CLINICAL TRIAL: NCT03083587
Title: Frequent Activity Snacks Breaks - Interrupting Sedentary Behaviour
Brief Title: Frequent Activity Snacks Breaks
Acronym: FABS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Baker Heart and Diabetes Institute (Other); Australian Catholic University (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Näslund, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016/1768
Record Dates: First submitted 2017-03-03; First posted 2017-03-20 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Insulin Resistance; Sedentary Lifestyle
MeSH Terms: conditions — Obesity; Insulin Resistance; Sedentary Behavior | interventions — Exercise; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (Active Comparator): Normal lifestyle. Subjects will undergo a muscle and fat biopsy at the start of the 4 w period and after. An oral glucose test at the start and after completion of the 4 week period. Physical activity and glucose will be monitored during the study period.
  Interventions: Behavioral: Normal lifestyle; Procedure: muscle and fat biopsy; Device: Continuous glucose monitoring; Device: Activity monitoring (ActivePal)
- Exercise intervention (Experimental): Followed by a 1 week normal run in period subjects will undergo a 3 min bout, every half hour between 8 am and 6 pm comprises of simple low-intensity exercise such as moderate walking about or climbing a flight of stairs over a 3-week period. Subjects will undergo a muscle and fat biopsy at the start of the 4 w period and after. An oral glucose test at the start and after completion of the 4 week period. Physical activity and glucose will be monitored during the study period.
  Interventions: Behavioral: Exercise; Procedure: muscle and fat biopsy; Device: Continuous glucose monitoring; Device: Activity monitoring (ActivePal)

INTERVENTIONS:
Behavioral: Normal lifestyle — Normal lifestyle
  Arms: No intervention
Behavioral: Exercise — Mild exercise 3 min every half hour
  Arms: Exercise intervention
Procedure: muscle and fat biopsy — Biopsy under local anesthesia
Device: Continuous glucose monitoring — Glucose concentrations during the study period
Device: Activity monitoring (ActivePal) — Objective measurements of standing and sitting time

SUMMARY:
There is a growing health burden in Sweden and Europe arising from the interrelated sequelae of metabolic disorders comprising impaired glucose tolerance (IGT), obesity and T2DM. Obesity and inactivity are the main drivers of IGT and T2DM and are responsible for up to 8% of health costs and 13% of deaths in Europe, with the risk of co-morbidities rising in parallel with increasing body weight. IGT and T2DM are the paradigm of inactivity-related disorders: the majority of people who have IGT or T2DM are overweight and inactive, with up to 80% being obese. A recent meta-analysis of 42 studies concluded that sedentary time was independently associated with a greater risk of T2D, all-cause mortality, cardiovascular disease incidence and mortality, and cancer incidence and mortality (breast, colon, colorectal, endometrial and epithelial ovarian cancers) (Ann Intern Med. 2015;162:123-32). A recent systematic review of trials published up to April 2014 identified 16 separate studies and concluded that there is considerable evidence of the positive effects of breaking up prolonged sitting time with light-intensity ambulatory physical activity and standing on postprandial metabolic parameters, including glucose, insulin and triglyceride levels (Med Sci Sports Exerc. 2015:47:2053-61). However, to date, all of the published experimental trials describing the beneficial effects of breaking up sitting time on metabolic risk markers have been restricted to acute exposure periods (1-5 days). We will perform a RCT intervention study, which examines the efficacy (clinically relevant responses) and practical implementation of low-impact training in sedentary obese individuals during the day.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle,
* BMI 30-40 kg/m2

Exclusion Criteria:

* Unable to read Swedish (for informed consent),
* anticoagulant therapy,
* unability to perform intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in metabolic health including insulin resistance | Change from baseline and 4 week intervention
  Oral glucose tolerance test including baseline glucose and insulin

SECONDARY OUTCOMES:
Changes at the molecular level in skeletal and fat muscle biopsies | Change from baseline and 4 week intervention
  insulin signalling cascade, the pathways that regulate protein synthesis and atrophy, as well as the content and function of mitochondria
Changes at the molecular level in skeletal and fat muscle biopsies | Change from baseline and 4 week intervention
  The pathways that regulate protein synthesis and atrophy
Changes at the molecular level in skeletal and fat muscle biopsies | Change from baseline and 4 week intervention
  Lipid, protein and metabolites
Changes in gene expression | Change from baseline and 4 week intervention
  RNA, mRNA, DNA methylation
Changes in physical activity | Change from baseline and 4 week intervention
  Objective measures of standing and sitting
Changes in plasma glucose | Change from baseline and 4 week intervention
  Continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Erik Naslund, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JAB, Savikj M, Sethi P, Platt S, Gabriel BM, Hawley JA, Dunstan D, Krook A, Zierath JR, Naslund E. Three weeks of interrupting sitting lowers fasting glucose and glycemic variability, but not glucose tolerance, in free-living women and men with obesity. Am J Physiol Endocrinol Metab. 2021 Aug 1;321(2):E203-E216. doi: 10.1152/ajpendo.00599.2020. Epub 2021 Jun 21. PMID 34151582